CLINICAL TRIAL: NCT02202447
Title: A Phase 1 Study of A Prostate-Specific Membrane Antigen Targeting-Tubulysin Conjugate EC1169 In Patients With Recurrent Metastatic, Castration-Resistant Prostate Cancer (MCRPC)
Brief Title: Phase 1 of EC1169 In Patients With Recurrent MCRPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC1169-01
Record Dates: First submitted 2014-07-21; First posted 2014-07-29 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: EC1169; prostate cancer; EC0652
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EC1169 (Experimental): PART A AND B: EC0652 is in development as a radioimaging agent for PSMA-expressing tumors. All patients receive a baseline 99mTc-EC0652 SPECT/CT scan for PSMA expression prior to Cycle 1 Day 1.
  PART A: EC1169 given as IV bolus QW on Weeks 1 and 2 of a 3 week cycle. Dose based on dose escalation plan starting with 0.2 mg/m2
  PART B: EC1169 cohort 1 - taxane naive mCRPC patients that have progressed while receiving (or subsequent to receiving) abiraterone and/or enzalutamide but must not have previously received taxane-based systemic chemotherapy for mCRPC (previous treatment with six cycles of docetaxel for metastatic castration-sensitive prostate cancer (mCSPC) is permissible).
  PART B: EC1169 cohort 2 - taxane exposed mCRPC patients who have progressed while receiving (or subsequent to receiving) abiraterone and/or enzalutamide and who have progressed subsequent to receiving > 2 cycles of a taxane-based regimen for mCRPC.
  Interventions: Drug: EC1169; Other: EC0652

INTERVENTIONS:
Drug: EC1169 — PART A: EC1169 - Dose dependent on cohort, IV (in the vein) on days 1 and 8 of each 21 day cycle for the QW schedule.
  PART B: EC1169 cohort 1 - taxane naive - Recommended Phase 2 dose, IV (in the vein) on days 1 and 8 of each 21 day cycle for the QW schedule.
  PART B: EC1169 cohort 2 - taxane exposed - Recommended Phase 2 dose, IV (in the vein) on days 1 and 8 of each 21 day cycle for the QW schedule.
Other: EC0652 — PART A AND B: EC0652 is in development as a radioimaging agent for PSMA-expressing tumors. All patients receive a baseline 99mTc-EC0652 SPECT/CT scan for PSMA expression prior to Cycle 1 Day 1.

SUMMARY:
The purpose of this study is to determine the safety of EC1169 and the best dose to use in humans in future studies. This study will also determine how EC1169 is distributed, broken down, passed and absorbed through your body and how quickly it is eliminated (leaves the body). All patients will receive EC1169.

As a secondary objective in Part A: To explore the relationships between baseline PSMA expression (tumor and patient level) as measured by 99mTc-EC0652 scans and the antitumor activity of EC1169.

As an exploratory objective in Part B: To assess EC0652 as a predictive biomarker for the efficacy of EC1169 by comparing PSMA-positive and PSMA-negative lesions for response.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, non-randomized, oncology study to conducted in 2 parts. Part A is a dose-escalation phase to determine the Recommended Phase 2 (RP2) dose and the following :

* Evaluate the administration of EC1169 QW on Weeks 1 and 2 of a 3-week schedule
* Evaluate the safety and pharmacokinetic profile of EC1169 and EC0652
* To assess preliminary efficacy results in patients with metastatic, castration-resistant prostate cancer (mCRPC) who have progressed on abiraterone and/or enzalutamide, and previously treated with a taxane.

The primary objective of Part B is to identify the radiographic progression-free survival (rPFS) in taxane-naïve and taxane-exposed PSMA-positive mCRPC patients receiving treatment with EC1169.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to sign an approved informed consent form (ICF).
* Patients must be ≥ 18 years of age.
* Patients must have histological, pathological and/or cytological confirmation of prostate cancer.
* Patients must have progressive, metastatic, castration-resistant prostate cancer (mCRPC) as defined below:
* Documented progressive metastatic CRPC will be based on at least one of the following criteria:

  * PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval and a minimum PSA of 2 ng/mL.
  * Soft-tissue progression defined as an increase ≥ 20% in the sum of the longest diameter (LD) of all target lesions based on the smallest sum LD since treatment started or the appearance of one or more new lesions.
  * Progression of bone disease (evaluable disease) or (new bone lesion(s)) by bone scan.
* Patients must have prior and/or ongoing androgen-deprivation therapy and a castrate level of serum testosterone (<50 ng/dL).
* Patients must have progressed on abiraterone and/or enzalutamide.
* Patients must have been previously treated with a taxane except in cases of contraindication (e.g. poor performance status, age or patient choice)
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must have at least one measurable lesion that can be followed for response assessment on baseline imaging obtained no more than 28 days prior to beginning study therapy. Baseline and follow up radiological disease assessment must include bone scans performed with either Technetium-99m labeled diphosphonates or Fluorine-18 sodium fluoride PET or PET/CT, as per the local standard of care for patients with prostate cancer.
* Patients with CNS metastases that are symptomatic must have received therapy (surgery, XRT, gamma knife) and be neurologically stable and off of steroids. The patient should be off steroids at least 14 days before pre-registration. Asymptomatic CNS metastatic disease without associated edema, shift, requirement for steroids or anti-seizure medications are eligible after discussion with the sponsor medical monitor. For patients with a history of CNS metastasis, baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast)
* Patients must have recovered (to baseline/stabilization) from prior therapy-associated acute toxicities.
* Patients with prior radiation therapy are eligible if they meet the following criteria:

  * Prior radiotherapy must be completed at least 4 weeks before patient begins study therapy.
  * Patient must have recovered from the acute toxic effects of the treatment before beginning study therapy.
* Patients must have adequate organ function:

  * Bone marrow reserve: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L. Platelets ≥ 100 x 109/L. Hemoglobin ≥ 9 g/dL.
  * Cardiac:
  * Left ventricular ejection fraction (LVEF) equal to or greater than the institutional lower limit of normal. LVEF must be evaluated within 28 days prior to beginning study therapy.
  * Cardiac Troponin I within normal limit.
* Hepatic: Total bilirubin ≤ 1.5 x the upper limit of normal (ULN). Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3.0 x ULN OR ≤ 5.0 x ULN for patients with liver metastases.
* Renal: Serum creatinine ≤ 1.5 x ULN, or for patients with serum creatinine > 1.5 ULN, creatinine clearance ≥ 50 mL/min.

Exclusion Criteria:

* More than 3 prior systemic anti-cancer therapies (e.g. cytotoxic agents, biologic agents) regimens for metastatic disease
* Previous treatment with Samarium-153 or Strontium-89.
* Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 28 days prior to beginning study therapy.
* Known hypersensitivity to the components of the study therapy or its analogs.
* Carcinomatous meningitis and/or symptomatic central nervous system (CNS) metastases.
* Malignancies that are expected to alter life expectancy or may interfere with disease assessment. Patients with adequately treated non-melanoma skin cancer and patients with prior history of malignancy who have been disease free for more than 3 years are eligible.
* Neuropathy CTCAE grade > 2
* QTc interval of > 480 ms.
* History of ischemic cardiac disease that has occurred within 6 months prior to study entry.
* Any other serious cardiac illness or medical conditions such as unstable angina, pulmonary embolism, or uncontrolled hypertension.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy.
* Active uncontrolled infections
* Known active Hepatitis B or C infections

Inclusion Criteria for Part B:

To qualify for enrollment, the following criteria must be met:

1. Patients must have the ability to understand, and have signed an approved ICF
2. Patients must be males ≥ 18 years of age
3. Patients must have histological, pathological and/or cytological confirmation of prostate cancer
4. Patients must have progressive mCRPC defined by meeting at least one of the following criteria:

   1. PSA progression defined as 25% increase over a baseline value of > 2 ng/ml with an increase in the absolute value of at least 2 ng/mL that is confirmed by another PSA level with a minimum of a 1-week interval. Baseline is defined as the PSA nadir level since commencing most recent prior therapy
   2. Soft-tissue progression defined as an increase ≥ 20% in the sum of the diameter (SOD; short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD, or the appearance of one or more new lesions, since the onset of the most recent prior therapy
   3. Progression of bone disease according to PCWG3 criteria
5. Patients must have a castrate level of serum testosterone (< 50 ng/dL)
6. For inclusion in Cohort 1, mCRPC patients must have progressed while receiving (or subsequent to receiving) abiraterone and/or enzalutamide but must not have previously received taxane-based systemic chemotherapy for mCRPC (previous treatment with six cycles of docetaxel for metastatic castration-sensitive prostate cancer (mCSPC) is permissible). NOTE: patients receiving fewer than 2 cycles of taxane based regimen due to intolerance are eligible for cohort 1.
7. For inclusion in Cohort 2, mCRPC patients must have progressed while receiving (or subsequent to receiving) abiraterone and/or enzalutamide and must have progressed subsequent to receiving ≥ 2 cycles of a taxane-based regimen for mCRPC.
8. Patients must have a ECOG performance status of 0 or 1
9. Patients must have at least one metastatic lesion that can be followed on baseline imaging obtained no more than 28 days prior to beginning study therapy. Baseline and follow up radiological disease assessments must include bone scans performed with 99mTc labelled diphosphonates
10. Patients with a history of CNS metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity. Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired. For patients with parenchymal CNS metastasis (or a history of CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast)
11. Patients must have recovered (to baseline/stabilization) from prior chemo- or radio-therapy and associated acute toxicities must have resolved to a NCI CTCAE v4 Grade 1 or less, with the exception of alopecia
12. Patients must have adequate organ function:

    a) Bone marrow reserve: ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 9 g/dL b) Cardiac: i) QTcF < 450 msec on at least 2 of 3 screening ECGs. On site determination of QTcF may be used for screening purposes ii) LVEF equal to or greater than the institutional lower limit of normal. LVEF must be evaluated within 7 to 10 days prior to beginning study therapy iii) Cardiac Troponin I within normal limit (as per local institution) c) Hepatic: Total bilirubin ≤ 1.5 x ULN, ALT, AST ≤ 3.0 x ULN OR ≤ 5.0 x ULN for patients with liver metastases d) Renal: Serum/plasma creatinine ≤ 1.5 x ULN, or for patients with serum/plasma creatinine > 1.5 ULN, creatinine clearance ≥ 50 mL/min

Exclusion Criteria for Part B:

The presence of any of the following will exclude the patient from the study:

1. Previous treatment with Samarium-153, Strontium-89, Rhenium-186 or Radium-223 within 6 months of starting (i.e., Cycle 1 Day 1) EC1169
2. Any systemic anti-cancer therapy (e.g., chemotherapy, immunotherapy or biological therapy (including monoclonal antibodies), or experimental anti-cancer therapy) within 28 days prior to beginning study therapy. Note: Ongoing castrating therapy with a GnRH agonist or antagonist is mandatory to assure a castrate level of serum testosterone <50 ng/dL, except in patients who have undergone an orchiectomy. Bisphosphonates or denosumab continuation is permissible (i.e., no change for 30 days prior to Cycle 1 Day 1). Patients who receive a dose of EC1169 under another Endocyte protocol do not need a washout period for EC1169
3. Known hypersensitivity to the components of the study therapy. (Please reference Section 1, Formulation of EC1169 and EC0652, in the respective Pharmacy Manuals)
4. Carcinomatous meningitis and/or symptomatic CNS metastases
5. Concurrent malignancies that are expected to alter life expectancy (e.g., NSCLC, etc.) or that may interfere with assessment of prostate cancer (e.g., lymphoma involving the periaortic nodes). Patients with adequately treated non-melanoma skin cancer or non-muscle invasive urothelial carcinoma, and patients with prior history of malignancy who have been disease-free for more than 5 years are eligible
6. Patients considered at risk for life-threatening QTc prolongation (i.e., personal or family history of Long QT syndrome, presence of implantable pacemaker, or implantable cardioverter defibrillator, etc.)
7. Use of the following medications within 6 months prior to EC1169 administration: amiodarone, disopyramide, dofetilide, dronedarone, flecanamide, ibutilide, quinidine, or sotalol
8. Any other serious cardiac illness or medical conditions such as unstable angina, pulmonary embolism, or uncontrolled hypertension
9. Known systemic infections including, but not limited to hepatitis B or C, or HIV

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
PART A: Maximum Tolerated Dose of EC1169 | Patients will be followed for an anticipated 21 days for occurence of DLTs
  Review to see if there are any (Dose Limiting Toxicities) seen in cycle 1.
PART B:To identify the radiographic progression-free survival (rPFS) in taxane-naïve and taxane-exposed PSMA-positive mCRPC | Patients will be followed until progression of disease or no longer clinically benefiting for an anticipated 27 weeks (9 cycles)
  To identify the radiographic progression-free survival (rPFS) in taxane-naïve and taxane-exposed PSMA-positive mCRPC patients receiving treatment with EC1169.

SECONDARY OUTCOMES:
PART A: Safety/adverse event review | Patients will be followed until progression of disease or unacceptable toxicity for an anticipated 12 weeks (4 cycles)
  Adverse Events reviewed weekly and at end of each cycle (every 21 days)
PART B: To evaluate time to Prostate Cancer Clinical Trials Working Group 3 (PCWG3)-defined NLCB (no longer clinically benefiting) | Patients will be followed until progression of disease or no longer clinically benefiting for an anticipated 27 weeks (9 cycles)
  To evaluate time to Prostate Cancer Clinical Trials Working Group 3 (PCWG3)-defined NLCB (no longer clinically benefiting)
PART B: To evaluate the median progression-free survival [defined as the time from C1D1 to an event (i.e., radiological or clinical progression or death)] for each cohort | Patients will be followed until progression of disease or no longer clinically benefiting for an anticipated 27 weeks (9 cycles)
  To evaluate the median progression-free survival [defined as the time from C1D1 to an event (i.e., radiological or clinical progression or death)] for each cohort

CONTACTS AND LOCATIONS:
Overall Officials: Alison Armour, MD, Study Director — Endocyte
Locations (6):
- United States (6):
  - Scottsdale Healthcare Clinical Trials at the Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Tulane Cancer Center, New Orleans, Louisiana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas